CLINICAL TRIAL: NCT06572436
Title: Evaluation of The Effect of Multimedia Information on Anxiety, Pain, Stress And Fear Levels Before Amniocentesıs And Chorıon Villus Sampling: A Randomized Controlled Study
Brief Title: Multımedia Information Before Amniocentesıs And Chorion Villus Sampling
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Akdeniz University (Other)
Responsible Party: Principal Investigator, Neriman Temel Aksu, Principal Investigator, Akdeniz University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: Akdenizpregnant
Record Dates: First submitted 2024-08-19; First posted 2024-08-27 (Actual); Last update posted 2024-08-27 (Actual); Status verified 2024-08

CONDITIONS: Amniocentesis; Chorionic Villus Sampling
Keywords: amniocentesis; anxiety; chorionic villus sampling; fear; multimedia information; pain; pregnant; stress
MeSH Terms: conditions — Anxiety Disorders; Pain

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Group (No Intervention): Pregnant women in the control group were not given multimedia information before amniocentesis and chorionic villus sampling, but were given brief verbal information about the procedure before amniocentesis and chorionic villus sampling.
- Multimedia information group (Experimental): Pregnant women in the study group were given multimedia information by watching a short video before amniocentesis and chorionic villus sampling. The multimedia information training consisted of a 5-minute video containing detailed amniocentesis and chorionic villus sampling application information. A 5-minute video was developed by the authors and used for research purposes only. The video was designed to provide pregnant women with a comprehensive overview of the amniocentesis and chorionic villus sampling procedure, its benefits, and potential risks, and included real-life images to depict all aspects of the procedure.
  Interventions: Behavioral: Multimedia information training

INTERVENTIONS:
Behavioral: Multimedia information training — The multimedia information training consisted of a 5-minute video containing detailed amniocentesis and chorionic villus sampling application information. A 5-minute video was developed by the authors and used for research purposes only. The video was designed to provide pregnant women with a comprehensive overview of the amniocentesis and chorionic villus sampling procedure, its benefits, and potential risks, and included real-life images to depict all aspects of the procedure.
  Arms: Multimedia information group

SUMMARY:
It is known that the anxiety levels of pregnant women are high before amniocentesis and chorionic villus sampling and it is often neglected. The aim of this study is to examine the effects of multimedia information given before invasive prenatal diagnostic tests such as amniocentesis and chorionic villus sampling on the anxiety, pain, stress and fear levels of pregnant women.

Pregnant women who are planned to undergo amniocentesis and chorionic villus sampling are included in this prospective randomized controlled study. 90 pregnant women are randomized into two groups as study (n=45) and control group (n=45). Pregnant women in the study group are educated with multimedia information before amniocentesis and chorionic villus sampling. Pregnant women in the control group are given brief verbal information about the procedure before amniocentesis and chorionic villus sampling. Anxiety, pain, stress and fear levels are assessed immediately before multimedia information and after amniocentesis and chorionic villus sampling.

DETAILED DESCRIPTION:
Prenatal invasive tests such as amniocentesis and chorionic villus sampling are performed to exclude or diagnose fetal chromosomal abnormalities. Most invasive diagnostic methods cause anxiety and fear in individuals, which can be a source of anxiety and depression in individuals. Although prenatal invasive tests are a simple and short procedure, they can result in serious discomfort and increased pain perception. Studies have determined that pregnant women have high anxiety levels before amniocentesis and chorionic villus sampling. Anxiety is the most common negative emotion associated with invasive procedures and is also a determinant of mood and pain sensation after the intervention. Concerns about pain and potential complications increase the anxiety experienced by pregnant women. There are very few studies addressing the psychological aspect associated with prenatal invasive tests. Studies have shown that women who are candidates for amniocentesis experience "state anxiety" and depressive symptoms.

Patient education reduces anxiety and worry. Various methods are used in patient education. Among these, verbal education, written material/brochures and multimedia-based education (videos, compact discs, digital versatile discs and the internet) are the most commonly used. The results regarding which method is more effective in patient education are unclear. Education given to pregnant women about the purposes, benefits, risks and limitations of amniocentesis can reduce anxiety and worry in pregnant women. Education increases pregnant women's awareness of the amniocentesis process and its results. Patients remember 20% of what is explained, 40% of what they read and 80% with multimedia education. Multimedia-based education has become more frequently used in patient education due to developments in the field of information technology. Multimedia education program is implemented through texts, shapes, sounds, animations and video clips to strengthen the learning activity of users. Multimedia not only increases the learning motivation of users, but also increases the learning activity. Multimedia education has no obstacles in terms of space or time. Therefore, if the equipment is ready, the user can directly access a specific topic in the program at any time and from anywhere.

It has been shown that a multimedia education program applied before radiologic imaging, endoscopy, colonoscopy, bronchoscopy, invasive cardiac approaches and arthroscopy does not cause cost loss and reduces patient anxiety. A multimedia education program applied before birth has been shown to increase pregnant women's knowledge and decision-making skills and reduce their anxiety. Multimedia education program before amniocentesis did not provide a significant reduction in the anxiety of pregnant women. In another study, a multimedia education program before amniocentesis; It has been shown to be an easy intervention that can be used to reduce the anxiety of pregnant women.

There are no sufficient studies investigating the effects of multimedia information given before amniocentesis on the anxiety levels of pregnant women. Furthermore, the effectiveness of multimedia information as an intervention to reduce anxiety before chorionic villus sampling has not been investigated. The aim of this study is to investigate the effects of a multimedia information video watched before invasive prenatal diagnostic tests such as amniocentesis and chorionic villus sampling on the anxiety, pain, stress and fear levels of pregnant women.

This prospective randomized controlled study is conducted on pregnant women who are scheduled to undergo amniocentesis and chorionic villus sampling by the responsible physician who applied to University Hospital Gynecology and Obstetrics Clinic, who did not have known cerebrovascular disease, who did not have morbid obesity or heart disease that would prevent the study, who did not have cognitive disorders that would prevent communication, who did not have a history of stroke or related effects, and who agreed to participate in the study. Pregnant women who had previously undergone amniocentesis and chorionic villus sampling and who did not agree to participate in the study are excluded from the study. Informed consent is obtained from the participants before amniocentesis and chorionic villus sampling procedures are performed. We used the CONSORT (Consolidated Standards of Reporting Trials) checklist while writing our report. The study is approved by the University Faculty of Medicine Clinical Research Ethics Committee.

The G-power v3.1 program (Universitat Kiel, Germany) is used to determine the sample size. Among the variables measured in the study, State-Trait Anxiety Inventory-I (STAI-I) is used as the basis for determining the sample size. When the effect size of the study is taken as f=0.50, α error level as 0.05, and power (1-β: error level) as 0.80, the total sample size is calculated as 90 pregnant women, including at least 45 controls. When the estimated individual loss rate during the study process is taken as 20%, it is planned to include at least 108 pregnant women in the study.

Initial evaluations are made for 108 pregnant women included in the study. Later, 12 pregnant women does not meet the study criteria and 6 pregnant women does not want to participate in the study and therefore dropped out. 90 pregnant women are randomized into two groups as study (n=45) and control group (n=45). They are randomized into two groups according to a number series consisting of 45 numbers prepared randomly between 1 and 90 through the randomization program random.org. The first of these number series is accepted as the study group and the second as the control group. Each pregnant woman included in the study is asked to draw one of the sealed envelopes containing the numbers between 1 and 90. The pregnant woman is assigned to the study or control group according to the number series containing the number drawn. The study is completed as study group (n=45) and control group (n=45). Since the studyis planned as single-blind, pregnant women are not informed about which study or control group they belonged to.

Pregnant women in the study group are given multimedia information by watching a short video before amniocentesis and chorionic villus sampling. Pregnant women in the control group are not given multimedia information before amniocentesis and chorionic villus sampling, but are given brief verbal information about the procedure before amniocentesis and chorionic villus sampling. The multimedia information training consist of a 5-minute video containing detailed amniocentesis and chorionic villus sampling application information. A 5-minute video is developed by the authors and used for research purposes only. The video is designed to provide pregnant women with a comprehensive overview of the amniocentesis and chorionic villus sampling procedure, its benefits, and potential risks, and included real-life images to depict all aspects of the procedure.

For the outcome measurements, anxiety level, pain, stress and fear levels are assessed. Anxiety level is assessed with STAI-I,II; pain, stress and fear levels are assessed with The Visual Analog Scale (VAS). After being included in the study, the initial anxiety, pain, stress and fear levels of the participants in both groups are assessed. Then, the participants in the study group watched the information video, while the pregnant women in the control group are given a standard verbal explanation. After the amniocentesis and chorionic villus sampling procedures, the second anxiety, pain, stress and fear levels of the participants in both groups are assessed.

The Personal Information Form is created as a result of a literature review on the subject in order to determine the number of gynecological examinations and birth information of the individuals participating in the sample. There are 27 questions in the Personal Information Form. Information that cannot be obtained from the pregnant woman will be obtained from the pregnant woman's relative or the pregnant woman's file; measurements such as body mass index calculation that cannot be accessed from the files will be made by the researcher.

State-Trait Anxiety Inventory-I and II (STAI-I-II) is translated into Turkish . STAI-I-II is used to measure temporary and permanent anxiety. These scales are four-point Likert type consisting of 20 items. While STAI-I describes an individual's feelings at a specific moment or under specific conditions, STAI-II describes how an individual feels regardless of the situation and conditions. The scale includes direct and indirect (reverse) statements. The total scores of the indirect (reverse) statements are subtracted from the total weighted scores obtained from the direct statements and a fixed value of 50 points is added for STAI-I and 35 points for STAI-II. The total score varies between 20 and 80, and scores of 45 and above are indicative of anxiety.

VAS is 10 cm long and is applied by marking a point corresponding to the intensity of pain, stress, and fear felt by the patient on a vertical or horizontal line with different names on both ends. The distance between the marked point and the lowest end of the line is measured in centimeters and the numerical value found indicates the intensity of pain, stress, and fear of the patient. 0 indicates no pain, stress, or fear, 1-3 indicates mild pain, stress, or fear, 4-6 indicates moderate pain, stress, or fear, and 7-10 indicates severe pain, stress, or fear. Verbal and numerical assessment scales, which are one-dimensional scales, are less sensitive and reliable in repeated measurements. The sensitivity and selectivity of the scale have been established and it is suitable for use. It will be used in the study to evaluate the level of anxiety and fear towards gynecological examination. Statistical analysis Data are analyzed using SPSS software (version 21.0; SPSS Inc, Chicago, IL). The one-sample Kolmogorov-Smirnov test is used to evaluate the distribution of variables before test selection. Descriptive statistics are expressed as frequency, mean, and standard deviation. Characteristics in the study and control groups are compared using the χ2 test for categorical variables and the Mann-Whitney U test for continuous variables. The Wilcoxon signed-rank test is used to compare within-group differences between baseline and post-intervention scores. The Mann-Whitney U test is used for between-group comparisons. Statistical significance is accepted as p<0.05. Effect sizes are calculated using the mean and standard deviation of the change scores for each group using GPower V.3.1.7 (University of Kiel, Kiel, Germany). The statistical significance level is P < .05.

ELIGIBILITY:
Inclusion Criteria:

pregnant women;

* who were scheduled to undergo amniocentesis and chorionic villus sampling by the responsible physician who applied to University Hospital Gynecology and Obstetrics Clinic,
* who did not have known cerebrovascular disease
* who did not have morbid obesity or heart disease that would prevent the study
* who did not have cognitive disorders that would prevent communication
* who did not have a history of stroke or related effects, and who agreed to participate in the study.

Exclusion Criteria:

* Pregnant women who had previously undergone amniocentesis and chorionic villus sampling and who did not agree to participate in the study

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2024-10-20 (Estimated); Primary Completion 2025-02-01 (Estimated); Study Completion 2025-04-01 (Estimated)

PRIMARY OUTCOMES:
Change of Anxiety Score | Change from Baseline Anxiety Score through study completion, an average of 1 hour
  State-Trait Anxiety Inventory-I and II (STAI-I-II) is used to measure temporary and permanent anxiety.. These scales are four-point Likert type consisting of 20 items. While the STAI-I describes an individual's feelings at a specific moment or under specific conditions, STAI-II describes how an individual feels regardless of the situation and conditions. The scale includes direct and indirect (reverse) statements. The total scores of the indirect (reverse) statements are subtracted from the total weighted scores obtained from the direct statements and a fixed value of 50 points is added for STAI-I and 35 points for STAI-II.
  After being included in the study, the initial anxiety levels of the participants in both groups are assessed. After the amniocentesis and chorionic villus sampling procedures, the second anxiety levels of the participants in both groups are assessed.
Change of Pain Score | Change from Baseline Pain Score through study completion, an average of 1 hour
  The Visual Analog Scale (VAS) was used as a one-dimensional scale for pain assessment. VAS is a self-administered, one-dimensional measure of pain intensity widely used in various adult populations. The VAS is a 10 cm long line in which participants mark the point they believe best represents the severity of pain. Always "0" means no pain, while "10" means excruciating pain.
  When asked, patients touch a point corresponding to their degree of pain, and this mark indicates the degree of pain on the scale. Higher scores indicate greater pain severity.
  After being included in the study, the initial pain levels of the participants in both groups are assessed. After the amniocentesis and chorionic villus sampling procedures, the second pain levels of the participants in both groups are assessed.
Change of Fear Score | Change from Baseline Fear Score through study completion, an average of 1 hour
  The Visual Analog Scale (VAS) was used as a one-dimensional scale for fear assessment. VAS is a self-administered, one-dimensional measure of pain intensity widely used in various adult populations. The VAS is a 10 cm long line in which participants mark the point they believe best represents the severity of fear. Always "0" means no pain, while "10" means excruciating fear.
  When asked, patients touch a point corresponding to their degree of fear, and this mark indicates the degree of fear on the scale. Higher scores indicate greater fear severity.
  After being included in the study, the initial fear levels of the participants in both groups are assessed. After the amniocentesis and chorionic villus sampling procedures, the second fear levels of the participants in both groups are assessed.
Change of Stress Score | Change from Baseline Stress Score through study completion, an average of 1 hour
  The Visual Analog Scale (VAS) was used as a one-dimensional scale for stress assessment. VAS is a self-administered, one-dimensional measure of stress intensity widely used in various adult populations. The VAS is a 10 cm long line in which participants mark the point they believe best represents the severity of stress. Always "0" means no pain, while "10" means excruciating stress.
  When asked, patients touch a point corresponding to their degree of stress, and this mark indicates the degree of stress on the scale. Higher scores indicate greater stress severity.
  After being included in the study, the initial stress levels of the participants in both groups are assessed. After the amniocentesis and chorionic villus sampling procedures, the second stress levels of the participants in both groups are assessed.

SECONDARY OUTCOMES:
Height in Meters | Initial assessment before amniocentesis and chorionic villus sampling .
  The height of all subjects in meters (m) will be noted before the surgery.
Weight in Kilograms | Initial assessment before amniocentesis and chorionic villus sampling .
  The weight of all subjects in kilograms (kg) will be noted before the surgery.
Body Mass Index (BMI) in kg/m^2 | Initial assessment before amniocentesis and chorionic villus sampling .
  Body Mass Index (BMI) will be calculated with the formula weight (kg)/height (m)^2.

CONTACTS AND LOCATIONS:
Overall Officials: Neriman Temel Aksu, Principal Investigator — Akdeniz University